CLINICAL TRIAL: NCT01358812
Title: Phase II Trial of FOLFOXIRI Plus Panitumumab as First-Line Treatment for Kras and Braf Wild-Type Metastatic Colorectal Cancer
Brief Title: FOLFOXIRI Plus Panitumumab In Kras and Braf Wild-Type Metastatic Colorectal Cancer
Acronym: TRIP
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Gruppo Oncologico del Nord-Ovest (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2934; 2009-014556-29 (EudraCT Number)
Record Dates: First submitted 2011-05-19; First posted 2011-05-24 (Estimated); Last update posted 2015-03-11 (Estimated); Status verified 2015-03

CONDITIONS: Metastatic Colo-rectal Cancer
Keywords: RAS Wild-Type; BRAF Wild-Type
MeSH Terms: conditions — Colonic Neoplasms | interventions — Panitumumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- FOLFOXIRI + Panitumumab (Experimental): PANITUMUMAB 6 mg/Kg i.v. over 1 hour followed by IRINOTECAN 150 mg/sqm i.v. over 1 hour followed by OXALIPLATIN 85 mg/sqm i.v. over 2 hours concomitantly with L-LV 200 mg/sqm over 2 hours followed by 5-FLUOROURACIL 2400 mg/sqm c.i. over 48 hours starting on day 1 repeated every 2 weeks.
  Interventions: Drug: FOLFOXIRI + Panitumumab

INTERVENTIONS:
Drug: FOLFOXIRI + Panitumumab — PANITUMUMAB 6 mg/Kg i.v. over 1 hour followed by IRINOTECAN 150 mg/sqm i.v. over 1 hour followed by OXALIPLATIN 85 mg/sqm i.v. over 2 hours concomitantly with L-LV 200 mg/sqm over 2 hours followed by 5-FLUOROURACIL* 2400 mg/sqm c.i. over 48 hours starting on day 1 repeated every 2 weeks.

SUMMARY:
The GONO-FOLFOXIRI regimen demonstrated higher activity and efficacy compared to FOLFIRI in a phase III trial. Panitumumab with oxaliplatin- or irinotecan-based doublets is feasible and associated with improved activity in KRAS codon 12-13 wild-type patients. BRAF and other RAS rare mutations have been suggested as additional potential biomarkers for anti-EGFR agents in metastatic colo-rectal cancer. The present study aims to demonstrate the feasibility and the activity of the first-line combination of the GONO-FOLFOXIRI regimen and Panitumumab in molecularly selected metastatic colo-rectal cancer patients.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed colorectal adenocarcinoma;
* Availability of formalin-fixed paraffin embedded tumor block from primary or metastasis;
* KRAS and BRAF wild-type status of primary colorectal cancer or related metastasis;
* Unresectable and measurable metastatic disease according to RECIST criteria;
* Male or female, aged >/= 18 years and </= 75 years;
* ECOG PS < 2 if aged < 71 years;
* ECOG PS = 0 if aged 71-75 years;
* Life expectancy of more than 3 months;
* Adequate haematological function: ANC ≥ 1.5 x 109/L; platelets ≥ 100 x 109/L, Hb ≥ 9 g/dL;
* Adequate liver function: serum bilirubin ≤ 1.5 x ULN; alkaline phosphatase and transaminases ≤ 2.5 x ULN (in case of liver metastases < 5 x ULN);
* Serum creatinine ≤ 1.5 x ULN;
* Previous adjuvant chemotherapy is allowed if more than 12 months have elapsed between the end of adjuvant therapy and first relapse;
* At least 6 weeks from prior radiotherapy and 4 weeks from surgery;
* Written informed consent to experimental treatment and pharmacogenomic analyses;
* Magnesium ≥ lower limit of normal;
* Calcium ≥ lower limit of normal.

Exclusion Criteria:

* Prior palliative chemotherapy;
* Prior treatment with EGFR inhibitors;
* Symptomatic peripheral neuropathy ≥ 2 grade NCIC-CTG criteria;
* Presence or history of CNS metastasis;
* Active uncontrolled infections; active disseminated intravascular coagulation;
* Past or current history of malignancies other than colorectal carcinoma, except for curatively treated basal and squamous cell carcinoma of the skin cancer or in situ carcinoma of the cervix;
* Clinically significant cardiovascular disease, for example cerebrovascular accidents (CVA) (≤ 6 months before treatment start), myocardial infarction (≤ 6 months before treatment start), unstable angina, NYHA ≥ grade 2 chronic heart failure (CHF), uncontrolled arrhythmia;
* Fertile women (< 2 years after last menstruation) and men of childbearing potential not willing to use effective means of contraception;
* Subject pregnant or breast feeding, or planning to become pregnant within 6 months after the end of treatment;
* History of interstitial lung disease e.g. pneumonitis or pulmonary fibrosis or evidence of interstitial lung disease on baseline chest CT scan.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2010-03; Primary Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Response Rate | Up to 3 years (objective response will be evaluated every 8 weeks)
  Response rate is defined as the fraction of treated patients who achieve a response as defined according to Response Evaluation Criteria in Solid Tumors (RECIST) criteria vers. 1.1.

SECONDARY OUTCOMES:
Progression Free Survival | Up to 3 years
  Progression free survival is defined as time from study entry until progression of disease (according to RECIST 1.1) or death from any cause. Patients who are alive without having progressed at the end of the study will be censored at their last radiological assessment.
Overall Survival | Up to 3 years
  Overall survival is defined as the time from study entry until death from any cause. Patients who are alive at the end of the study will be censored at that point.
Safety Profile | Up to 3 years
  Safety Profile is based on the collection of all the adverse events occurring during the study graded by NCI-CTC criteria.
Secondary Radical Surgery on Metastases | Up to 3 years
  Secondary Radical Surgery on Metastases is defined as microscopically margin-free complete surgical removal of all residual disease performed during treatment or after its completion allowed by tumoral shrinkage and or desappearance of one or more lesions.
Analyses of Potential Predictive Factors | Up to 3 years
  Exploratory analyses of potential predictive factors and surrogate markers of treatment activity or efficacy.

CONTACTS AND LOCATIONS:
Overall Officials: Alfredo Falcone, MD, Principal Investigator — Polo Oncologico Area Vasta Nord-Ovest
Locations (10):
- Italy (10):
  - P.O. Zona Aretina - Ospedale S. Donato Di Arezzo, Arezzo
  - Istituto Nazionale Per La Ricerca Sul Cancro, Genova
  - IRCCS Ospedale San Raffaele, Milan
  - Asl Olbia - Uo Oncologia Ospedale San Giovanni Di Dio, Olbia
  - Istituto Oncologico Veneto (IOV), Padua
  - Polo Oncologico Area Vasta Nord-Ovest, Pisa
  - Universita' Campus Bio-Medico Di Roma, Roma
  - Asl Di Sassari - Ospedale S.S. Annunziata -U.O. Oncologia Medica, Sassari
  - Ausl 7 Di Siena, Siena
  - A.O. Universitaria S.Maria Della Misericordia Di Udine, Udine

REFERENCES:
- [Background] Falcone A, Ricci S, Brunetti I, Pfanner E, Allegrini G, Barbara C, Crino L, Benedetti G, Evangelista W, Fanchini L, Cortesi E, Picone V, Vitello S, Chiara S, Granetto C, Porcile G, Fioretto L, Orlandini C, Andreuccetti M, Masi G; Gruppo Oncologico Nord Ovest. Phase III trial of infusional fluorouracil, leucovorin, oxaliplatin, and irinotecan (FOLFOXIRI) compared with infusional fluorouracil, leucovorin, and irinotecan (FOLFIRI) as first-line treatment for metastatic colorectal cancer: the Gruppo Oncologico Nord Ovest. J Clin Oncol. 2007 May 1;25(13):1670-6. doi: 10.1200/JCO.2006.09.0928. PMID 17470860
- [Background] Douillard JY, Siena S, Cassidy J, Tabernero J, Burkes R, Barugel M, Humblet Y, Bodoky G, Cunningham D, Jassem J, Rivera F, Kocakova I, Ruff P, Blasinska-Morawiec M, Smakal M, Canon JL, Rother M, Oliner KS, Wolf M, Gansert J. Randomized, phase III trial of panitumumab with infusional fluorouracil, leucovorin, and oxaliplatin (FOLFOX4) versus FOLFOX4 alone as first-line treatment in patients with previously untreated metastatic colorectal cancer: the PRIME study. J Clin Oncol. 2010 Nov 1;28(31):4697-705. doi: 10.1200/JCO.2009.27.4860. Epub 2010 Oct 4. PMID 20921465
- [Background] Peeters M, Price TJ, Cervantes A, Sobrero AF, Ducreux M, Hotko Y, Andre T, Chan E, Lordick F, Punt CJ, Strickland AH, Wilson G, Ciuleanu TE, Roman L, Van Cutsem E, Tzekova V, Collins S, Oliner KS, Rong A, Gansert J. Randomized phase III study of panitumumab with fluorouracil, leucovorin, and irinotecan (FOLFIRI) compared with FOLFIRI alone as second-line treatment in patients with metastatic colorectal cancer. J Clin Oncol. 2010 Nov 1;28(31):4706-13. doi: 10.1200/JCO.2009.27.6055. Epub 2010 Oct 4. PMID 20921462
- [Background] De Roock W, Claes B, Bernasconi D, De Schutter J, Biesmans B, Fountzilas G, Kalogeras KT, Kotoula V, Papamichael D, Laurent-Puig P, Penault-Llorca F, Rougier P, Vincenzi B, Santini D, Tonini G, Cappuzzo F, Frattini M, Molinari F, Saletti P, De Dosso S, Martini M, Bardelli A, Siena S, Sartore-Bianchi A, Tabernero J, Macarulla T, Di Fiore F, Gangloff AO, Ciardiello F, Pfeiffer P, Qvortrup C, Hansen TP, Van Cutsem E, Piessevaux H, Lambrechts D, Delorenzi M, Tejpar S. Effects of KRAS, BRAF, NRAS, and PIK3CA mutations on the efficacy of cetuximab plus chemotherapy in chemotherapy-refractory metastatic colorectal cancer: a retrospective consortium analysis. Lancet Oncol. 2010 Aug;11(8):753-62. doi: 10.1016/S1470-2045(10)70130-3. Epub 2010 Jul 8. PMID 20619739